CLINICAL TRIAL: NCT04802278
Title: Gestational Immunity for Transfer
Acronym: GIFT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: National University of Singapore (Other); Agency for Science, Technology and Research (Other)
Responsible Party: Sponsor
Other Study IDs: 2021/00095
Record Dates: First submitted 2021-03-15; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Covid19; Breastfeeding; Vaccine Exposure Via Breast Milk
MeSH Terms: conditions — COVID-19; Breast Feeding | interventions — COVID-19 Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Babies born to mothers convalescent from antenatal COVID-19
- Babies born to healthy mothers
- Vaccinated mothers: Lactating mothers who received COVID-19 vaccination
  Interventions: Biological: COVID-19 vaccine

INTERVENTIONS:
Biological: COVID-19 vaccine — Any COVID-19 vaccine
  Groups: Vaccinated mothers

SUMMARY:
This is a study prospective cohort study at an urban academic centre, with two parts:

1. Health outcomes, and maternally transferred antibodies, in babies born to mothers who had antenatal COVID-19 and convalesced before delivery, followed up until 12 months of age
2. Safety and protective properties of breast milk after lactating women are vaccinated against COVID-19

DETAILED DESCRIPTION:
This proposal aims to provide a multi-faceted approach to study how immunity may be transferred - both transplacentally and through breastfeeding, from mother to child, in the context of COVID-19.

We first recruit all babies delivered to mothers convalescent from antenatal COVID-19, to 1) follow up their growth and development, and 2) study the protective effects of antibodies transferred from mother to child transplacentally during pregnancy, as well as postnatally through breastfeeding. We compare these to a cohort of healthy controls whose mothers did not have COVID-19 during pregnancy.

Next, we compare the protective effects of antibodies transferred during breastfeeding from mother to child after lactating mothers are vaccinated against COVID-19, to that of natural infection. We also study the safety of breastfeeding after vaccination by looking for vaccine components in the breast milk.

ELIGIBILITY:
Inclusion Criteria:

Lives in Singapore

Exclusion Criteria:

Prematurity Congenital abnormalities Primary immunodeficiencies Autoimmune disorders

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — For group 3; only lactating women recruited
Study Population: Part 1 of study - infants Part 2 of study - lactating women
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Transplacentally transferred antibodies | From birth to 12 months of age
  Binding and neutralising immunoglobulin G specific to SARS-CoV-2 spike and receptor-binding domain
Antibodies transferred through breast milk (convalescent mothers) | From birth to 6 months of age
  Binding and neutralising immunoglobulin A specific to SARS-CoV-2 spike and receptor-binding domain
Antibodies transferred through breast milk (vaccinated mothers) | From just before vaccination, to 6 weeks after vaccination
  Binding and neutralising immunoglobulin A specific to SARS-CoV-2 spike and receptor-binding domain

SECONDARY OUTCOMES:
General health | From birth to 12 months of age
  Growth and development of infants

CONTACTS AND LOCATIONS:
Locations (1):
- National University Hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gu Y, Low JM, Tan JSY, Ng MSF, Ng LFP, Shunmuganathan B, Gupta R, MacAry PA, Amin Z, Lee LY, Lian D, Shek LP, Zhong Y, Wang LW. Immune and pathophysiologic profiling of antenatal coronavirus disease 2019 in the GIFT cohort: A Singaporean case-control study. Front Pediatr. 2022 Sep 15;10:949756. doi: 10.3389/fped.2022.949756. eCollection 2022. PMID 36186648
- [Derived] Low JM, Lee LY, Ng YPM, Zhong Y, Amin Z. Breastfeeding Mother and Child Clinical Outcomes After COVID-19 Vaccination. J Hum Lact. 2022 Feb;38(1):37-42. doi: 10.1177/08903344211056522. Epub 2021 Oct 29. PMID 34713745